CLINICAL TRIAL: NCT01894516
Title: Randomized, Double-blind, Placebo-controlled, Multicenter, Phase IIb Dose Finding Study of GLPG0634 Administered for 24 Weeks as Monotherapy to Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate (MTX) Alone
Brief Title: Dose-finding Study of GLPG0634 as Monotherapy in Active Rheumatoid Arthritis (RA) Participants (DARWIN2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-204 (DARWIN2)
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants received GLPG0634 matching placebo capsules, orally, once daily (QD) during Weeks 1 to 12 and GLPG0634 100 milligram (mg) QD during Weeks 13 to 24.
  Interventions: Drug: Placebo
- GLPG0634 50 mg QD (Experimental): Participants received GLPG0634 50 mg capsules, orally, QD during Weeks 1 to 12. Participants who were responders (having at least 20% improvement on TJC68 and SJC66) remained on 50 mg QD while nonresponders were re-randomized to 100 mg QD during Weeks 13 to 24.
  Interventions: Drug: GLPG0634
- GLPG0634 100 mg QD (Experimental): Participants received GLPG0634 100 mg capsules, orally, QD during Weeks 1 to 24.
  Interventions: Drug: GLPG0634
- GLPG0634 200 mg QD (Experimental): Participants received GLPG0634 200 mg capsules, orally, QD during Weeks 1 to 24.
  Interventions: Drug: GLPG0634

INTERVENTIONS:
Drug: GLPG0634 — GLPG0634 capsules.
  Arms: GLPG0634 100 mg QD; GLPG0634 200 mg QD; GLPG0634 50 mg QD
Drug: Placebo — Placebo capsules.
  Arms: Placebo

SUMMARY:
* Participants suffering from active rheumatoid arthritis who had an inadequate response to methotrexate were evaluated for improvement of disease activity (efficacy) when taking GLPG0634 as monotherapy (3 different doses - 50 milligram (mg), 100 mg and 200 mg once daily) or matching placebo for 24 weeks.
* During the course of the study, patients were also examined for any side effects that could occur (safety and tolerability), and the amount of GLPG0634 present in the blood (Pharmacokinetics) as well as the effects of GLPG0634 on disease- and mechanism of action-related parameters in the blood (Pharmacodynamics) were determined. Also, the effects of different doses of GLPG0634 administration on participants' disability, fatigue and quality of life were evaluated.

DETAILED DESCRIPTION:
* Treatment duration was 24 weeks in total.
* However, at Week 12, all participants on placebo and the participants on the 50 mg dose who had not achieved 20% improvement in swollen joint count (SJC66) and tender joint count (TJC68) were assigned (automatically via interactive web response system (IWRS)) to 100 mg once daily (QD) in a blinded fashion and continued treatment until Week 24.
* Participants in the other groups maintained their randomized treatment until Week 24.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects who are ≥18 years of age on the day of signing informed consent,
* have a diagnosis of RA since at least 6 months and meeting the 2010 ACR/EULAR criteria of RA and ACR functional class I-III,
* have ≥6 swollen joints (from a 66-joint count) and

  ≥8 tender joints (from a 68-joint count) at Screening and at Baseline,
* Screening serum c-reactive protein ≥ 0.7 x upper limit of laboratory normal range (ULN),
* have shown an inadequate response in terms of either lack of efficacy or toxicity to MTX,
* have agreed to be washed out from MTX for a period of at least 4 weeks before or during the Screening period.

Exclusion Criteria:

* current therapy with any non-biological disease modifying anti-rheumatic drug (DMARD), with the exception of antimalarials, which must be at a stable dose for at least 12 weeks prior to Screening,
* current or previous RA treatment with a biologic DMARD, with the exception of biologic DMARDs: administered in a single clinical study setting, and; more than 6 months prior to Screening (12 months for rituximab or other B cell depleting agents), and; where the biologic DMARD was effective, and if discontinued, this should not be due to lack of efficacy,
* previous treatment at any time with a cytotoxic agent, other than MTX, before Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2013-10-08 (Actual); Primary Completion 2015-03-05 (Actual); Study Completion 2015-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (82):
- United States (21):
  - Artho Care, Arthritis Care & Research P.C., Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Research PLLC, Mesa, Arizona
  - Arizona Arthritis Rheum Res, Phoenix, Arizona
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - C.V. Mehta MD Medical Corp., Hemet, California
  - Center for Innovative Therapy Division of Rheumatology, UCSD, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - Infosphere Clinical Research, Inc., West Hills, California
  - Lovelace Scientific Resources, Venice, Florida
  - Arthritis Center of North GA, Gainesville, Georgia
  - The Arthritis Center, Springfield, Illinois
  - Klein and Associates MD, Hagerstown, Maryland
  - Private practice, Lansing, Michigan
  - Arthritis Center of Reno, Reno, Nevada
  - New Jersey Physicians, LLC, Clifton, New Jersey
  - Health research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center Clin Research, Duncansville, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - Austin Rheumatology Research PA, Austin, Texas
  - Pioneer Research Solutions Inc, Houston, Texas
- Argentina (3):
  - Centro de Investigaciones Medicas Lanus, Lanús
  - Instituto Centralizado de Asistencia e investigacion Clinica Integral, Rosario
  - Centro Médico Privado de Reumatología, San Miguel de Tucumán
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown
  - Princess Alexandra Hospital, Woolloongabba
- Rheumazentrum Favoriten, Vienna, Austria
- Bulgaria (2):
  - "Multiprofile Hospital for Active Treatment - Kaspela" LTD, Plovdiv
  - Clinic of Rheumatology MHAT, Sofia
- Chile (2):
  - Hospital Regional "Guillermo Grant Benavente", Concepción
  - Private Office, Temuco
- Colombia (6):
  - Fundación del Caribe para la Investigación Biomédica BIOS, Barranquilla
  - Centro Integral de Reumatologia SAS, Bogotá
  - Cirei Sas, Bogotá
  - Idearg S.A.S., Bogotá
  - Medicity S.A.S., Bucaramanga
  - Preventive Care Ltda, Chía
- Germany (2):
  - Schlossparkklinik - Akad. Lehrkrankenhaus Charite, Berlin
  - Schwerpunktpraxis fuer Rheumatologie, Hamburg
- Guatemala (3):
  - Clinica Médica Especializada en Medicina Interna, Guatemala City
  - Reuma S.A., Guatemala City
  - Reuma-Centro, Guatemala City
- Hungary (4):
  - DRC, Balatonfüred
  - Qualiclinic Ltd, Budapest
  - Revita Clinic, Budapest
  - Csolnoky Ferenc County Hospital, Veszprém
- Latvia (2):
  - L. Atikes doktorats, Liepāja
  - "Bruninieku" Polyclinic, Riga
- Mexico (6):
  - Arké Estudios Clínicos S.A. de C.V., México
  - Centro Medico Dalinde, México
  - Clinstile, S.A. de C.V., México
  - Mexico Centre for Clinical Research, México
  - Hospital Universitario, Monterrey
  - Hospital de Especialidades, Oaxaca City
- IMSP Institutul de Cardiologie, Chisinau, Moldova
- New Zealand (2):
  - North Shore hospital, Auckland
  - Timaru Rheumatology Studies, Timaru
- Poland (10):
  - Silesiana Centrum Medyczne, Bytom
  - Centrum Kliniczno, Elblag
  - Medica Pro Familia Sp. z o.o. S.K.A., Katowice
  - Nowomed, Krakow
  - Nzoz "Dobry Lekarz", Krakow
  - NZOZ Przychodnia Lekarska "Eskulap", Skierniewice
  - NZOZ Medicus Bonus, Środa Wielkopolska
  - AMED Medical Center, Warsaw
  - Ars Rheumatica Sp. Z.o.o., Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
- Romania (4):
  - Ianuli Med Consult SRL, Bucharest
  - Sana Medical Center, Bucharest
  - Spitalul Clinic Sfanta Maria, Bucharest
  - Emergency County Hospital, Galati
- Russia (3):
  - Orenburg State Medical Academy, Orenburg
  - GUZ "Regional Clinical Hospital", Saratov
  - Vladimir Reg Clin Hosp, Vladimir
- Spain (3):
  - Hospital General Elche, Elche
  - Consorci Sanitari Parc Tauli, Sabadell
  - CICEC S.L.P Hospital Ntra.Sra.de la Esperanza, Santiago de Compostela
- Ukraine (5):
  - V. Gusak Institute of Urgent and Recovery Surgery, Donetsk
  - City Hospital #8, Kharkiv
  - Municipal Hospital, Kherson
  - Central Outpatient Hospital of Deanyanskyy Distric, Kiev
  - Regional Clinical Hospital, Vinnytsia

REFERENCES:
- [Derived] Balsa A, Wassenberg S, Tanaka Y, Tournadre A, Orzechowski HD, Rajendran V, Lendl U, Stiers PJ, Watson C, Caporali R, Galloway J, Verschueren P. Effect of Filgotinib on Body Mass Index (BMI) and Effect of Baseline BMI on the Efficacy and Safety of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Dec;10(6):1555-1574. doi: 10.1007/s40744-023-00599-1. Epub 2023 Sep 25. PMID 37747626
- [Derived] Combe B, Besuyen R, Gomez-Centeno A, Matsubara T, Sancho Jimenez JJ, Yin Z, Buch MH. Geographic Analysis of the Safety and Efficacy of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Feb;10(1):35-51. doi: 10.1007/s40744-022-00494-1. Epub 2022 Oct 7. PMID 36205910
- [Derived] Tarrant JM, Galien R, Li W, Goyal L, Pan Y, Hawtin R, Zhang W, Van der Aa A, Taylor PC. Filgotinib, a JAK1 Inhibitor, Modulates Disease-Related Biomarkers in Rheumatoid Arthritis: Results from Two Randomized, Controlled Phase 2b Trials. Rheumatol Ther. 2020 Mar;7(1):173-190. doi: 10.1007/s40744-019-00192-5. Epub 2020 Jan 7. PMID 31912462
- [Derived] Kavanaugh A, Kremer J, Ponce L, Cseuz R, Reshetko OV, Stanislavchuk M, Greenwald M, Van der Aa A, Vanhoutte F, Tasset C, Harrison P. Filgotinib (GLPG0634/GS-6034), an oral selective JAK1 inhibitor, is effective as monotherapy in patients with active rheumatoid arthritis: results from a randomised, dose-finding study (DARWIN 2). Ann Rheum Dis. 2017 Jun;76(6):1009-1019. doi: 10.1136/annrheumdis-2016-210105. Epub 2016 Dec 19. PMID 27993828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Latin America, Europe, United States, and New Zealand. The first participant was screened on 08 October 2013. The last study visit occurred on 29 May 2015.
Pre-assignment Details: A total of 625 participants were screened of which 287 participants were randomized into the study and only 283 participants were treated.
Groups:
- GLPG0634 50 mg QD: Participants received GLPG0634 50 mg capsules, orally, QD during Weeks 1 to 12. Participants who were responders (having at least 20 percent [%] improvement on TJC68 and SJC66) remained on 50 mg QD while nonresponders were re-randomized to 100 mg QD during Weeks 13 to 24.
Period: Period 1 (Baseline up to Week 12)
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Started | 72 | 72 | 70 | 69
Completed | 65 | 67 | 67 | 66
Not Completed | 7 | 5 | 3 | 3
Not completed — Other | 0 | 1 | 1 | 0
Not completed — Adverse event and treatment failure | 2 | 0 | 0 | 0
Not completed — Non compliance with the study medication | 1 | 1 | 0 | 0
Not completed — Treatment failure | 0 | 0 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 2
Period: Period 2 (Week 13 to Week 24)
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Started | 0 (All participants from Placebo moved to 100 mg QD (65 participants) group.) | 52 (Nonresponders from 50 mg QD group moved to 100 mg QD group (15 participants).) | 147 (Nonresponders from Placebo(65 participants) and 50 mg QD (15 participants) moved to 100 mg QD group.) | 66
Completed | 0 | 50 | 142 | 65
Not Completed | 0 | 2 | 5 | 1
Not completed — Adverse Event | 0 | 2 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were randomized and received at least one dose of study medication.
Groups:
- Placebo: Participants received GLPG0634 matching placebo capsules, orally, QD during Weeks 1 to 12 and GLPG0634 100 mg QD during Weeks 13 to 24.
- Total: Total of all reporting groups
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD | Total
Number analyzed (Participants) | 72 | 72 | 70 | 69 | 283
Age, Continuous [Mean (Full Range); unit: years] | 51.5 [20 to 77] | 52.1 [18 to 79] | 52.8 [22 to 78] | 51.8 [25 to 79] | 52.1 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 62 | 53 | 60 | 231
  Male | 16 | 10 | 17 | 9 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 23 | 25 | 25 | 98
  Not Hispanic or Latino | 47 | 49 | 45 | 44 | 185
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 53 | 53 | 53 | 54 | 213
  More than one race | 17 | 17 | 16 | 15 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Rheumatoid Arthritis (RA) duration [Mean (Full Range); unit: years] | 9.46 [0.7 to 28.9] | 8.63 [0.5 to 23.4] | 8.57 [0.5 to 33.7] | 8.68 [0.5 to 49.6] | 8.84 [0.5 to 49.6]
C-reactive protein (CRP) at Baseline [Mean (Full Range); unit: milligram per liter (mg/L)] | 35.26 [1 to 175] | 24.67 [1 to 162.9] | 25.55 [1.6 to 244.1] | 23.16 [1 to 91.3] | 27.21 [1.0 to 244.1]
Corrected tender joint count based on 68 joints (TJC68) at Baseline [Mean (Full Range); unit: joint count] — 68 joints were assessed for tenderness and joints are classified as tender/not tender giving a total possible tender joint count score of 0 to 68.
  joint count | 25.226 [8 to 63] | 25.58 [9 to 64] | 27.195 [8 to 65] | 26.242 [8 to 65.94] | 26.051 [8 to 65.94]
Corrected swollen joint count based on 66 joints (SJC66) at Baseline [Mean (Full Range); unit: joint count] — 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66.
  joint count | 15.98 [7 to 38] | 16.969 [7 to 48] | 18.653 [6 to 56] | 15.74 [6 to 46] | 16.834 [6 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an American College of Rheumatology (ACR) 20 Response at Week 12
Description: The American College of Rheumatology (ACR) response is a measurement of improvement in multiple disease assessment criteria. The ACR20 response is defined as: 1) ≥ 20% improvement from baseline in SJC66, and 2) ≥ 20% improvement from baseline in tender TJC68, and 3) ≥ 20% improvement from baseline in at least 3 of the following 5 items: 1. Pain visual analog scale (VAS) (taken from the Health Assessment Questionnaire - Disability Index [HAQ-DI]), 2. Patient's Global Assessment of Disease Activity VAS, 3. Physician's Global Assessment of Disease Activity VAS, 4. Total HAQ-DI score, and 5. CRP. Non-responder imputation was used (ie, to impute a missing response, the participant was assumed to be a non-responder).
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all participants in the safety population who had post-randomization data for at least one efficacy parameter.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received GLPG0634 matching placebo capsules, orally, QD during Weeks 1 to 12 and GLPG0634 100 mg, QD during Weeks 13 to 24.
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 72 | 72 | 70 | 69
percentage of participants | 29.2 | 66.7 | 65.7 | 72.5
Statistical Analysis 1: Comparison: Placebo vs GLPG0634 50 mg QD; Pairwise comparisons of each group vs. the placebo group using a logistic regression model with factors treatment group, geographical region, and prior use of biologics; Test type: Superiority; p < 0.0001, Regression, Logistic — P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 37.5, 95% CI 2-sided [22.4 to 52.6]
Statistical Analysis 2: Comparison: Placebo vs GLPG0634 100 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 36.5, 95% CI 2-sided [21.3 to 51.8]
Statistical Analysis 3: Comparison: Placebo vs GLPG0634 200 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — P-value has been corrected for multiplicity according to Hommel's closed-testing method; Difference in percentage rates = 43.3, 95% CI 2-sided [28.4 to 58.2]

2. Secondary Outcome: Percentage of Participants Achieving an ACR20 Response at Week 24
Description: ACR20 response was defined as: 1) ≥ 20% improvement from baseline in SJC66, and 2) ≥ 20% improvement from baseline in TJC68, and 3) ≥ 20% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI), 2. Patient's Global Assessment of Disease Activity VAS, 3. Physician's Global Assessment of Disease Activity VAS, 4. Total HAQ-DI score, and 5. CRP. Non-responder imputation was used.
Time Frame: Week 24
Population: All patients from the ITT population who were randomized to a GLPG0634 arm. The data for participants switching from placebo to GLPG0634 100 mg at Week 12 were not in scope for this analysis and were not reported.
Measure: Number; unit: percentage of participants
Arm/Group | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 72 | 70 | 69
percentage of participants | 56.9 | 78.6 | 66.7

3. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response at Weeks 1, 2, 4, 8, 12, and 24
Description: ACR50 response was defined as: 1) ≥ 50% improvement from baseline in SJC66, and 2) ≥ 50% improvement from baseline in TJC68, and 3) ≥ 50% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI) 2. Patient's Global Assessment of Disease Activity VAS 3. Physician's Global Assessment of Disease Activity VAS 4. Total HAQ-DI score 5. CRP. Non-responder imputation was used. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: ITT population. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 72 | 72 | 70 | 69
percentage of participants
  Week 1 | 1.4 | 1.4 | 10 | 7.2
  Week 2 | 4.2 | 5.6 | 7.1 | 21.7
  Week 4 | 4.2 | 15.3 | 18.6 | 23.2
  Week 8 | 5.6 | 16.7 | 25.7 | 31.9
  Week 12 | 11.1 | 34.7 | 37.1 | 43.5
  Week 24: number analyzed (Participants) | 0 | 72 | 70 | 69
  Week 24 |  | 33.3 | 38.6 | 44.9

4. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response at Weeks 1, 2, 4, 8, 12, and 24
Description: ACR70 response: 1) ≥ 70% improvement from baseline in SJC66, and 2) ≥ 70% improvement from baseline in TJC68, and 3) ≥ 70% improvement from baseline in at least 3 of the following 5 items: 1. Pain VAS (taken from the HAQ-DI), 2. Patient's Global Assessment of Disease Activity VAS, 3. Physician's Global Assessment of Disease Activity VAS, 4. Total HAQ-DI score, and 5. CRP. Non-responder imputation was used. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: ITT population with available data were analyzed. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 72 | 72 | 70 | 69
percentage of participants
  Week 1 | 0 | 0 | 1.4 | 1.4
  Week 2 | 2.8 | 1.4 | 1.4 | 4.3
  Week 4 | 1.4 | 8.3 | 5.7 | 11.6
  Week 8 | 2.8 | 6.9 | 11.4 | 17.4
  Week 12 | 2.8 | 8.3 | 18.6 | 13
  Week 24: number analyzed (Participants) | 0 | 72 | 70 | 69
  Week 24 |  | 19.4 | 25.7 | 24.6

5. Secondary Outcome: ACR N% Improvement (ACR-N) Response at Weeks 1, 2, 4, 8, 12, and 24
Description: The ACR-N is the smallest percentage improvement in swollen and tender joints and the median of the remaining 5 core parameters, and is expected to be more sensitive to change than the ACR20, ACR50 or ACR70. It is a number varying between 0 and 100, with higher numbers indicating less severity of symptoms. Last observation carried forward (LOCF) algorithm was used (ie, to impute a missing value, the last preceding nonmissing value was used). All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percentage of improvement
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 72 | 72 | 70 | 69
percentage of improvement
  Week 1 | 6.79 (1.34) | 11.66 (1.641) | 12.84 (2.291) | 16.8 (2.346)
  Week 2 | 10.79 (1.917) | 17.11 (2.362) | 16.06 (2.261) | 27.01 (2.776)
  Week 4 | 12.03 (2.058) | 25 (2.852) | 24.06 (2.898) | 32.21 (3.172)
  Week 8 | 13.35 (2.24) | 30.46 (2.986) | 32.66 (3.154) | 39.24 (3.375)
  Week 12 | 16.28 (2.723) | 35.03 (3.178) | 38.35 (3.533) | 41 (3.477)
  Week 24: number analyzed (Participants) | 0 | 72 | 70 | 69
  Week 24 |  | 38.75 (3.748) | 46.32 (3.295) | 46.78 (3.648)

6. Secondary Outcome: Percentage of Participants With Disease Activity Score 28 Joints Corrected for CRP (DAS28 (CRP)) European League Against Rheumatism (EULAR) Response at Weeks 1, 2, 4, 8, 12, and 24
Description: DAS28 (CRP) was categorized into EULAR response categories (none, moderate, good) as follows: None = Actual DAS28 (CRP) ≤ 3.2, > 3.2 to ≤ 5.1, or > 5.1 AND Improvement in DAS28 (CRP) from baseline ≤ 6.0 or > 0.6 to ≤ 1.2; Moderate = Actual DAS28 (CRP) ≤ 3.2 AND Improvement in DAS28 (CRP) from baseline > 0.6 to ≤ 1.2, Actual DAS28 (CRP) > 3.2 to ≤ 5.1 or > 5.1 AND Improvement in DAS28 (CRP) from baseline > 1.2, or Actual DAS28 (CRP) > 3.2 to ≤ 5.1 AND Improvement in DAS28 (CRP) from baseline > 0.6 to ≤ 1.2; Good = Actual DAS28 (CRP) ≤ 3.2 AND Improvement in DAS28 (CRP) from baseline > 1.2. LOCF algorithm was used. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 72 | 72 | 70 | 69
percentage of participants
  Week 1: None | 72 | 57 | 63 | 49
  Week 1: Moderate | 26 | 40 | 31 | 43
  Week 1: Good | 1 | 3 | 6 | 7
  Week 2: None | 67 | 44 | 47 | 26
  Week 2: Moderate | 31 | 49 | 46 | 64
  Week 2: Good | 3 | 7 | 7 | 10
  Week 4: None | 58 | 38 | 39 | 22
  Week 4: Moderate | 35 | 47 | 46 | 55
  Week 4: Good | 7 | 15 | 16 | 23
  Week 8: None | 54 | 36 | 24 | 12
  Week 8: Moderate | 36 | 39 | 54 | 54
  Week 8: Good | 10 | 25 | 21 | 35
  Week 12: None | 49 | 31 | 20 | 14
  Week 12: Moderate | 38 | 46 | 53 | 41
  Week 12: Good | 14 | 24 | 27 | 45
  Week 24: None: number analyzed (Participants) | 0 | 72 | 70 | 69
  Week 24: None |  | 28 | 9 | 10
  Week 24: Moderate: number analyzed (Participants) | 0 | 72 | 70 | 69
  Week 24: Moderate |  | 36 | 41 | 43
  Week 24: Good: number analyzed (Participants) | 0 | 72 | 70 | 69
  Week 24: Good |  | 36 | 50 | 46

7. Secondary Outcome: Percentage of Participants Achieving ACR/EULAR Remission at Weeks 2, 4, 8, 12, and 24
Description: A participant's disease activity status can be defined as being in remission when scores on the TJC28, SJC28, CRP (actual value in mg/dL) and Patient Global Assessment of Disease Activity (cm) are all ≤ 1. Non-responder imputation was used. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Weeks 4, 8, 12, and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 72 | 72 | 70 | 69
percentage of participants
  Week 4 | 0 | 1.4 | 0 | 1.4
  Week 8 | 0 | 0 | 0 | 7.2
  Week 12 | 1.4 | 1.4 | 4.3 | 4.3
  Week 24: number analyzed (Participants) | 0 | 72 | 70 | 69
  Week 24 |  | 8.3 | 8.6 | 8.7

8. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 1, 2, 4, 8, 12, and 24
Description: The SDAI is the numerical sum of 5 outcome parameters: TJC28, SJC28, Patient Global Assessment of Disease Activity (in cm), Physician's Global Assessment of Disease Activity (in cm), and CRP (mg/dL). The SDAI was categorized as follows: • High disease activity: SDAI > 26 • Moderate disease activity: 11 to 26 • Low disease activity: 3.3 to 11 • Remission: ≤ 3.3. LOCF algorithm was used. The SDAI total score ranges from 0 to approximately 86. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 71 | 70 | 70 | 68
units on a scale
  Baseline | 45.73 (1.4789) | 43.77 (1.5609) | 46.608 (1.6538) | 44.139 (1.5079)
  Change at Week 1 | -7.45 (1.5528) | 9.596 (1.2567) | -10.886 (1.6511) | -14.349 (1.4346)
  Change at Week 2 | -10.022 (1.371) | -12.194 (1.5982) | -13.172 (1.6209) | -18.27 (1.6934)
  Change at Week 4 | -10.927 (1.7771) | -17.57 (1.7653) | -18.862 (1.8073) | -21.288 (1.6619)
  Change at Week 8 | -12.452 (1.7748) | -20.144 (1.9425) | -23.119 (1.8041) | -25.556 (1.6949)
  Change at Week 12 | -12.574 (1.984) | -21.413 (1.7953) | -25.269 (1.9856) | -26.499 (1.7534)
  Change at Week 24: number analyzed (Participants) | 0 | 70 | 70 | 68
  Change at Week 24 |  | -23.16 (1.9364) | -30.983 (1.7732) | -29.564 (1.8583)

9. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 1, 2, 4, 8, 12, and 24
Description: The CDAI is the SDAI modified to exclude CRP and is the sum of the 4 outcome parameters: TJC28, SJC28, Patient Global Assessment of Disease Activity (in cm), and Physician's Global Assessment of Disease Activity (in cm). The CDAI was be categorized as follows: • High disease activity: > 22 • Moderate disease activity: 10 to 22 • Mild disease activity: 2.8 to 10 • Remission: ≤ 2.8. LOCF algorithm was used. The CDAI total score ranges from 0 to approximately 76. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, and 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 71 | 70 | 70 | 68
units on a scale
  Baseline | 42.168 (1.3272) | 41.438 (1.4777) | 44.052 (1.5383) | 41.869 (1.423)
  Change at Week 1 | -6.867 (1.4538) | -9.226 (1.1545) | -9.853 (1.5591) | -13.148 (1.4085)
  Change at Week 2 | -9.861 (1.1909) | -11.803 (1.5275) | -12.306 (1.5618) | -16.999 (1.702)
  Change at Week 4 | -10.743 (1.7184) | -16.701 (1.7003) | -17.654 (1.6987) | -20.044 (1.6396)
  Change at Week 8 | -12.071 (1.6982) | -19.087 (1.8583) | -21.703 (1.7491) | -24.228 (1.6479)
  Change at Week 12 | 11.696 (1.8752) | -21.019 (1.7168) | -24.044 (1.9665) | -25.071 (1.742)
  Change at Week 24: number analyzed (Participants) | 0 | 70 | 70 | 68
  Change at Week 24 |  | -22.278 (1.8637) | -29.502 (1.6928) | -28.102 (1.818)

10. Secondary Outcome: Change From Baseline in Quality of Life Using the Functional Assessment of Chronic Illness Therapy (FACIT) at Weeks 4, 12, and 24
Description: FACIT-Fatigue scale is a 13-item questionnaire, each scored on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated that are scored reversely), the greater the fatigue. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score), with a higher score indicating a better quality of life. LOCF algorithm was used. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: ITT population with available data were analyzed. Participants who switched treatment at Week 12 were handled as if they discontinued at Week 12. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 71 | 70 | 70 | 69
units on a scale
  Baseline | 25.1 (1.12) | 25.1 (1.28) | 24.8 (1.13) | 24.8 (1.16)
  Change at Week 4 | 1.4 (1.14) | 7.2 (1.3) | 7.2 (1.26) | 8.5 (1.3)
  Change at Week 12 | 3.9 (1.23) | 9.5 (1.43) | 10.2 (1.21) | 11.2 (1.44)
  Change at Week 24: number analyzed (Participants) | 0 | 70 | 70 | 69
  Change at Week 24 |  | 10 (1.43) | 11.3 (1.2) | 13.7 (1.38)

11. Secondary Outcome: Change From Baseline in Quality of Life Using the Short Form-36 (SF-36) Scores at Weeks 4, 12, and 24
Description: The SF-36 is a 36-item questionnaire measuring 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status. Two summary scale scores were computed based on weighted combinations of the 8 domain scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). LOCF algorithm was used. All placebo participants switched to GLPG0634 treatment at Week 12 and were not included in the analysis of Week 24.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
Number analyzed (Participants) | 71 | 70 | 70 | 69
units on a scale
  PCS at Baseline | 31.1 (0.6988) | 31.05 (0.816) | 30.946 (0.7631) | 31.804 (0.8965)
  PCS Change at Week 4 | 2.1 (0.72) | 5.7 (1.04) | 5.1 (0.92) | 6.8 (0.92)
  PCS Change at Week 12 | 3 (0.89) | 7.1 (1.11) | 7.8 (1.04) | 8.6 (1.09)
  PCS Change at Week 24: number analyzed (Participants) | 0 | 70 | 70 | 69
  PCS Change at Week 24 |  | 6.9 (1.16) | 10 (1.17) | 9.7 (1.09)
  MCS at Baseline | 40.525 (1.3053) | 42.793 (1.3247) | 41.185 (1.2347) | 42.613 (1.1674)
  MCS at Week 4 | 2.1 (1.1) | 3.6 (1.09) | 5.3 (1.04) | 3.9 (1.16)
  MCS at Week 12 | 2.7 (1.04) | 4.9 (1.18) | 6.9 (1.04) | 6.8 (1.33)
  MCS at Week 24: number analyzed (Participants) | 0 | 70 | 70 | 69
  MCS at Week 24 |  | 5.1 (1.27) | 7.7 (1.16) | 8.5 (1.12)

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average exposure: 161.0 days)
Description: Nonresponders from 50 mg QD (15 participants) moved to 100 mg QD group for Week 13 to 24.
Arm/Group | Placebo | GLPG0634 50 mg QD | GLPG0634 100 mg QD | GLPG0634 200 mg QD
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72 | 0/85 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/72 | 2/72 | 3/85 | 3/69
Other Adverse Events (participants affected / at risk) | 9/72 | 14/72 | 21/85 | 16/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | GLPG0634 50 mg QD (N=72) | GLPG0634 100 mg QD (N=85) | GLPG0634 200 mg QD (N=69)
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | GLPG0634 50 mg QD (N=72) | GLPG0634 100 mg QD (N=85) | GLPG0634 200 mg QD (N=69)
Hypertension (Vascular disorders) | 4 | 3 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 4
Headache (Nervous system disorders) | 1 | 4 | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 4 | 5 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 3 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT01894516/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT01894516/SAP_001.pdf